CLINICAL TRIAL: NCT00580177
Title: Prolene Hernia System, Lichtenstein Mesh, and Plug-and-Patch for Primary Inguinal Hernia Repair - Three Year Outcome of a Prospective Randomised Controlled Trial
Brief Title: PHS, Lichtenstein Mesh, and PerFixPlug for Primary Inguinal Hernia Repair - 3 Years Results
Acronym: BOOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Jan Dalenbäck Associate Professor, Frolunda Specialist Hospital, Univeristy of Gothenburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSS BOOP
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Hernia, Inguinal
Keywords: Inguinal hernia; Randomized controlled trial; Surgery; Complications; Surgical mesh
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- L (Active Comparator): The Lichtenstein procedure for repair of inguinal hernia (Single On-lay patch)
  Interventions: Procedure: Lichtenstein mesh
- P (Active Comparator): The well-konown PerFixPlug technique for inguinal hernia repair.
  Interventions: Procedure: PerFix Plug®
- PHS (Active Comparator): The well-known Prolene Hernia System method for inguinal hernia repair.
  Interventions: Procedure: Prolene® Hernia System

INTERVENTIONS:
Procedure: Lichtenstein mesh — The different techniques are compared and evaluated according to primary and secondary objectives.
  Other Names: Inguinal hernioplasty (surgical repair of inguinal hernia)
  Arms: L
Procedure: PerFix Plug® — The different techniques are compared and evaluated according to primary and secondary objectives.
  Other Names: Inguinal hernioplasty (surgical repair of inguinal hernia)
  Arms: P
Procedure: Prolene® Hernia System — The different techniques are compared and evaluated according to primary and secondary objectives.
  Other Names: Inguinal hernioplasty (surgical repair of inguinal hernia)
  Arms: PHS

SUMMARY:
Three different techniques for the surgical repair of groin hernias are compared. Focus has been set on operation times, time to full return of functional abilities like walking in stairs etc, and if any technique has more complications than the others. Three years results are presented in the study.

DETAILED DESCRIPTION:
Dissection requirements differ between various methods for inguinal hernia repair, which may effect operation times, pain response and possibly recovery time. The objectives of this study were to establish if any differences concerning these aspects could be detected after three principally different techniques for primary inguinal hernia repair.

472 men between 30 and 75 years with primary inguinal hernias were included in a prospective controlled study and randomised to Lichtenstein mesh (L), PerFix Plug® (P) or the Prolene® Hernia System (PHS) procedure. All patients were seen and data were collected after 2 weeks, 3 months, 1 year, and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-75 years
* Men
* Primary inguinal hernia
* ASA I-III

Exclusion Criteria:

* > 75 years
* Females
* ASA IV
* Previous ipsi-lateral hernia surgery
* Drug or alchol abuse
* Severe illness

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2000-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Time until full functional recovery | 2 weeks, 3 months, 1 year, 3 years
Operation time | Registered after completion of surgery
Pain after operation measured on a VAS-scale and amount of consumed analgesics | Day 1-14, 3 months, 1 year, 3 years after surgery

SECONDARY OUTCOMES:
Complication rate | 2 weeks, 3 months, 1 year, 3 years
Aptness for beeing performed under local anaesthesia | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Dalenbäck, Ass. Prof., Principal Investigator — Frolunda Specialist Hospital, University of Gothenburg; Jan A Dalenbäck, Ass. Prof., Study Director — Frolunda Specialist Hospital, University of Gothenburg
Locations (1):
- Frolunda Specialist Hoospital/University of Gothenburg, Lundby Hospital, Molndals Hospital/Sahlgrens University Hospital, Gothenburg, Vastra Gotalandsregionen, Sweden